CLINICAL TRIAL: NCT01005628
Title: Velcade - Regulatory Post Marketing Surveillance (PMS)
Brief Title: Bortezomib (Velcade) - Regulatory Post Marketing Surveillance (PMS)
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR012958; bortezomib PMS (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Multiple Myeloma
Keywords: Bortezomib postmarketing surveillance; Korea bortezomib PMS
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001: bortezomib Injection into a vein 1.3 mg/m2 twice a week for 21 days
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — Injection into a vein 1.3 mg/m2 twice a week for 21 days

SUMMARY:
After the KFDA (Korea Food and Drug Administration) approval of a new drug, an annual report of the drug's safety and efficacy data must be reported to the Health Authority in 6 years. In this Observational study, we will investigate the basic demographic, medical history, concomitant drug use, as well as dosing information of multiple myeloma patients using bortezomib (Velcade).

DETAILED DESCRIPTION:
After the KFDA approval of a new drug, an annual report of the drug's safety and efficacy data must be reported to the Health Authority in 6 years. In this Observational study, we will investigate the basic demographic, medical history, concomitant drug use, as well as dosing information of multiple myeloma patients using bortezomib (Velcade). We will collect the response rate according to the EMBT (European Group for Blood and Marrow Transplant; a non-profit organization based in the Netherlands that promotes the transplantation of haemopoietic stem cells from all donor sources and donor types and related basic and clinical research, education, standardization, quality control, and accreditation for transplant procedures) or IMWG (the International Myeloma Working Group) criteria and the adverse events to assess the efficacy and safety. Observational Study - No investigational drug administered

ELIGIBILITY:
Inclusion Criteria:

* Patients who are newly prescribed bortezomib injection for the treatment of multiple myeloma

Exclusion Criteria:

* Patients who are hypersensitive to the bortezomib or any component of the bortezomib or with a history of the hypersensitivity
* Patients with severe hepatic impairment
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are newly prescribed bortezomib injection for the treatment of multiple myeloma in Korea
Sampling Method: Non-Probability Sample
Enrollment: 1121 (Actual)
Dates: Start 2006-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The data on AE (Adverse event) incidence, such as whether AEs occurred, types of AEs, and incidence of AEs by type | every cycles or every 3 weeks

SECONDARY OUTCOMES:
The overall response rate (complete remission rate+partal remission rate) will be measured according to the EBMT or IMWG criteria. | every cycle or every 3 weeks and end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.
Locations (1):
- Seoul, South Korea